CLINICAL TRIAL: NCT00000761
Title: Phase I/II Study of Recombinant Human Interferon-gamma (rIFN-gamma) in HIV-Infected Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 211; 11188 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Interferon-gamma, Recombinant; Acquired Immunodeficiency Syndrome; AIDS-Related Complex
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — interferon gamma-1b

INTERVENTIONS:
Drug: Interferon gamma-1b

SUMMARY:
PRIMARY: To determine the safety and toxicity of recombinant interferon gamma-1b ( rIFN-gamma ) in HIV-infected children receiving ongoing zidovudine ( AZT ) or didanosine ( ddI ) therapy. To document HIV-associated defects in neutrophil and/or monocyte function that are improved with rIFN-gamma.

SECONDARY: To determine whether a change in CD4 cell count occurs and to assess virologic status and effects on AZT and ddI pharmacokinetics.

It is likely that infants and children severely immunocompromised by HIV infection would respond to immunomodulators that augment different portions of the host defense system. Interferon-gamma has been shown to benefit children with severely compromised nonspecific immunity and may thus be of benefit to those with HIV infection.

DETAILED DESCRIPTION:
It is likely that infants and children severely immunocompromised by HIV infection would respond to immunomodulators that augment different portions of the host defense system. Interferon-gamma has been shown to benefit children with severely compromised nonspecific immunity and may thus be of benefit to those with HIV infection.

Patients are treated with subcutaneous rIFN-gamma 3 times a week for 24 weeks and are then followed for an additional 12 weeks.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required:

* AZT or ddI therapy.
* PCP prophylaxis.

Allowed:

* Antipyretics.
* Antiemetics.
* Antihistamines.
* Decongestants.
* Skin creams and lotions.
* Immunizations according to current recommendations.

Patients must have:

* Class P-2 symptomatic HIV infection.
* Ongoing AZT or ddI therapy of 6 months or longer duration.

Exclusion Criteria

Concurrent Medication:

Excluded:

* Antiretroviral therapy other than AZT or ddI.
* Chemotherapy for active malignancy.
* Amphotericin B for systemic fungal infections.

Patients with the following prior conditions are excluded:

* History of congestive heart failure or arrhythmias.
* History of congenital heart disease.
* History of seizure disorder requiring anticonvulsant medication. (NOTE:

History of uncomplicated febrile seizures does not exclude.)

Prior Medication:

Excluded within 8 weeks prior to study entry:

* Immunomodulators other than IVIG.

Prior Treatment:

Excluded:

* Red blood cell transfusion within 4 weeks prior to study entry.

Required:

* Ongoing AZT or ddI therapy of 6 weeks or longer duration.
* Ongoing PCP prophylaxis for more than 6 weeks duration.

Ongoing alcohol or drug use.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20
Dates: Study Completion 1997-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: WT Shearer, Study Chair; SL Abramson, Study Chair; MW Kline, Study Chair
Locations (2):
- United States (2):
  - The Children's Hosp. of Philadelphia IMPAACT CRS, Philadelphia, Pennsylvania
  - Texas Children's Hosp. CRS, Houston, Texas

REFERENCES:
- [Background] Kline MW, Fletcher CV, Douglas SD, Fenton T, Shearer WT. Recombinant human interferon-gamma (rIFN-gamma) treatment of HIV-infected children. Conf Retroviruses Opportunistic Infect. 1997 Jan 22-26;4th:143 (abstract no 424)
- [Background] Shearer WT, Kline MW, Abramson SL, Fenton T, Starr SE, Douglas SD. Recombinant human gamma interferon in human immunodeficiency virus-infected children: safety, CD4(+)-lymphocyte count, viral load, and neutrophil function (AIDS Clinical Trials Group Protocol 211). Clin Diagn Lab Immunol. 1999 May;6(3):311-5. doi: 10.1128/CDLI.6.3.311-315.1999. PMID 10225828